CLINICAL TRIAL: NCT05689502
Title: intenSive UpPer Extremity Recovery Program for Chronic Stroke (SUPER)
Acronym: SUPER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sean Savitz, Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-22-0774
Record Dates: First submitted 2023-01-09; First posted 2023-01-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Chronic Stroke
Keywords: Rehabilitation; Arm recovery; High intensity therapy; Occupational therapy; Physical therapy
MeSH Terms: interventions — Therapeutics

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Device: Treatment

INTERVENTIONS:
Device: Treatment — Subjects will participate in 6 hours of therapy a day, 5 days a week, for 3 consecutive weeks. These sessions will include 2 hours of occupational therapy, 2 hours of physical therapy, and 2 hours of guided individual work. Some of these sessions will be in a group setting. The therapy sessions will be individualized to the subject's personal goals and will focus on improving the function of the arm most affected by the stroke. Sessions may include electrical stimulation of the muscles, if it is determined to be safe. At the end of each week, the therapists will recommend exercises for the subjects to continue to work on at home on the weekend.

SUMMARY:
The purpose of this study is to Investigate the feasibility of a high-quality, high-dose, high-intensity upper extremity therapy program and to assess the treatment effects of a high-quality, high-dose, high-intensity upper extremity therapy program on functional outcomes, motor impairment, and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Single qualifying stroke event as confirmed by CT or MRI
* At least 6 months post stroke
* Fugl-Meyer upper extremity (UE) score of 20-45
* Able to follow written instructions
* Able to tolerate 6 hours of therapy a day

Exclusion Criteria:

* Prior arm injury impacting available passive or active range of motion or significant arm pain with movement
* Active drug or alcohol abuse
* Diagnosed with advanced dementia
* Pre-stroke baseline mRS>3
* History of clinically significant ischemic or hemorrhagic stroke resulting in prior arm weakness in the same territory as the index stroke
* Medical instability assessed by the treating stroke physician to participate to the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in integrity of the contralateral corticospinal tract fibers as assessed by the MRI with Diffusion Tensor Imaging (DTI) evaluation | Baseline(1 week prior to intervention),within 1 week after intervention
Change in functional arm movements as assessed by the Fugl Meyer-Upper Extremity Assessment | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This is a 66 item questionnaire and each is scored from 0(cannot perform)-2(performs fully) a higher score indicating better outcome
Change in functional gross and fine motor coordination as assessed by the Action Research Arm Test (ARAT) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This test has 4 subscales and each measures grasp, grip, pinch and gross movement.
  The Grasp subscale has 6 questions and is scored from 0-18, higher score indicating better outcome The Grip subscale has 4 items and is scored from 0-12, higher score indicating better outcome The Pinch subscale has 6 items and is scored from 0-18, higher score indicating better outcome The Gross movement subscale has 3 items and is scored from 0-9, higher score indicating better outcome

SECONDARY OUTCOMES:
Change in degree of disability as assessed by the Modified Rankin Scale (mRS) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  mRS is a 6 point disability scale with possible scores from 0(no disability) to 5(disability requiring constant care) a higher score indicating more disability
Change in performance in activities of daily living as assessed by the Barthel Index (BI) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This is a scoring technique that measures performance in ten activities of daily living including feeding, wheelchair to bed transfers, grooming ,chair to toilet transfers, walking, using stairs, dressing, and continence of bowels and bladder. This is a 10 item questionnaire and is scored from 0-100, a higher score indicating higher level of independence.
Change in fatigue as assessed by the Neurological Fatigue Index (NFI) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This is a 12 item questionnaire and each is scored on a 4 point Likert scale from 0(strongly disagree) to 3(strongly agree)
Change in anxiety as assessed by the Hospital Anxiety and Depression Scale (HADS) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This consists of 7 questions and each is scored from 0(not at all) to 3(most of the time) for a maximum score of 21, a higher number indicating more anxiety
Change in depression as assessed by the Hospital Anxiety and Depression Scale (HADS) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This consists of 7 questions and each is scored from 0(not at all) to 3(most of the time) for a maximum score of 21, a higher number indicating more depression
Change in functional ability of the hemiplegic arm and hand to perform meaningful tasks as assessed by the Chedoke Arm and Hand Inventory (CAHAI) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This contains 13 tasks and each is scored from 7(complete independence) to 1(total assistance) for a maximum score of 91, a higher number indicating better outcome
Change in difficulty to care for the affected arm as assessed by the Arm Activity Measure A | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This consists of 8 questions and each is scored from 0(no difficulty) to 4(unable to do activity) for a maximum score of 32 a higher number indicating worse outcome
Change in difficulty in completing functional tasks with the affected arm as assessed by the Arm Activity Measure B | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  This consists of 13 questions and each is scored from 0(no difficulty) to 4(unable to do activity) for a maximum score of 52 a higher number indicating worse outcome
Change in cognitive impairment as measured by the Montreal Cognitive Assessment (MoCA) | Baseline (1 week prior to the intervention), within 1 week after the intervention, 6 weeks after intervention, 6 months after intervention
  Total score on the Montreal Cognitive Assessment (MoCA) range from 0 to 30, with a higher score indicating a better outcome

OTHER OUTCOMES:
Number of participants that had a positive perception of the intervention as indicated by the semi structured interview | Once between 6 week and 6 month assessments.
Number of participants that had functional arm improvement after the intervention as indicated by the semi structured interview | Once between 6 week and 6 month assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Savitz, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No